CLINICAL TRIAL: NCT03769961
Title: Ataxia in Essential Tremor: Describing the Differences Between Disease Process and Treatment Effect (ATAX)
Brief Title: Ataxia in Essential Tremor: Describing the Differences Between Disease Process and Treatment Effect
Acronym: ATAX
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amie Hiller, MD, Associate Professor, Oregon Health and Science University
Other Study IDs: 18608
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Essential Tremor; Deep Brain Stimulation; Ataxia; Cerebellar Diseases
Keywords: essential tremor; dbs
MeSH Terms: conditions — Essential Tremor; Ataxia; Cerebellar Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ET (DBS-, Ataxia+): Essential Tremor without DBS with Ataxia on examination
  Interventions: Other: No intervention
- ET (DBS-, Ataxia-): Essential Tremor without DBS and without Ataxia on examination
  Interventions: Other: No intervention
- ET (DBS+, Ataxia+): Essential Tremor with DBS with Ataxia on examination
  Interventions: Other: No intervention
- ET (DBS+, Ataxia-): Essential Tremor with DBS without Ataxia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No interventions - Observational study

SUMMARY:
The proposed study aims to characterize ataxia occurring in essential tremor and essential tremor with DBS.

DETAILED DESCRIPTION:
Objectives: In recent years, there has been a growing amount of evidence tying Essential Tremor (ET) to cerebellar dysfunction. This has been clinically observed, demonstrated through specific gait measures of ataxia (often involving tandem gait), and confirmed through Positron emission tomography (PET) imaging. Deep Brain stimulation for ET has become a widely utilized therapeutic intervention for patients, and the bilateral thalamic ventralis intermedius (VIM) is most commonly implanted. However, it has been noted that in some patients gait ataxia significantly worsens post-op. This initially was thought to be a result of disease progression, but recent studies have in fact shown that this is a DBS related phenomenon.

Methods: Participants will have two visits to either the Portland VA or Oregon Health & Science University (OHSU). At each visit, several assessments of balance, tremor, gait and balance, and DBS settings will be made. The gait and balance assessments will be performed by a unblinded and a blinded rater.

ELIGIBILITY:
Inclusion Criteria:

* Essential Tremor diagnosis at least 3 years duration
* Absence of other neurological signes (such as dystonia, ataxia, or Parkinsonism)
* Patients must be able to walk 2 minutes unassisted.
* Patients must be able to understand and consent to be in the study.

Exclusion Criteria:

* Patients who have had changes in DBS settings within the last 3 months.
* Patients who have had no initial improvement or response to DBS.
* ET medication changes in the last month.
* Actively abusing alcohol.
* A neurologic diagnosis other than ET that in the investigator's opinion could affect gait and/or balance.
* Atypical tremor disorder including by not limited to tremor due to multiple sclerosis, medication-induced tremor, Parkinson's disease, or parkinsonian syndrome.
* Dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Essential Tremor participants with and without ataxia
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Ataxia Differences between DBS and no DBS | Visit 2 (after DBS has been turned off for 3-10 days)
  Compare the Scale of the Assessment and Rating of Ataxia (SARA) total score between DBS and no DBS participants with essential tremor. This 8-item scale rates gait (0-8 points), stance (0-6 points), sitting (0-4 points), speech disturbance (0-6 points), finger chase (0-4 points), nose-finger test (0-4 points), fast alternating hand movements (0-4 points), and heel-shin slide (0-4 points). Motor activists of the four extremities (items 5-8) assessments are performed bilaterally, mean values to obtain a total score. Cumulative score ranges from 0 (no ataxia) to 40 (most severe ataxia).

SECONDARY OUTCOMES:
Balance Confidence | Visit 2 (after DBS has been turned off for 3-10 days)
  The Activities-Specific Balance Confidence Scale (ABC) is a subjective measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness. The ABC scale is a 16-item self-report measure in which participants rate their balance confidence on a 0-100 scale (0 = 0 no confidence, 100 = 100 complete confidence). Overall score is calculated by adding item scores and dividing by the total number of items.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Post data entry and verification, data and specimens will be de-identified (no 18 HIPAA identifiers and age aggregated for those > 89 years old) and transferred to the Neurological Disorder Repository (MIRB # 3129). This repository is maintained at the Portland VA Health Care System. Verification of the coded data set creation and the absence of the identifiers will be created and retained in the study files. The research coordinator will be responsible for the creation and verification process. The key to the code will be maintained by the study and will not be released to the repository. The recipient investigator must present the data use agreement, documentation of an Institutional Review Boar (IRB) approved protocol and Informed Conset Form (ICF) allowing the release of the identifiable specimens/data, or the release of coded specimens/data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Board. Requestors will be required to sign a data access agreement.
URL: https://www.portland.va.gov/research/

REFERENCES:
- [Background] Ramirez-Zamora A, Boggs H, Pilitsis JG. Reduction in DBS frequency improves balance difficulties after thalamic DBS for essential tremor. J Neurol Sci. 2016 Aug 15;367:122-7. doi: 10.1016/j.jns.2016.06.001. Epub 2016 Jun 2. PMID 27423573
- [Result] Nazzaro JM, Lyons KE, Pahwa R. Deep brain stimulation for essential tremor. Handb Clin Neurol. 2013;116:155-66. doi: 10.1016/B978-0-444-53497-2.00013-9. PMID 24112892
- [Result] Kronenbuerger M, Konczak J, Ziegler W, Buderath P, Frank B, Coenen VA, Kiening K, Reinacher P, Noth J, Timmann D. Balance and motor speech impairment in essential tremor. Cerebellum. 2009 Sep;8(3):389-98. doi: 10.1007/s12311-009-0111-y. Epub 2009 May 19. PMID 19452239
- [Result] Fasano A, Herzog J, Raethjen J, Rose FE, Muthuraman M, Volkmann J, Falk D, Elble R, Deuschl G. Gait ataxia in essential tremor is differentially modulated by thalamic stimulation. Brain. 2010 Dec;133(Pt 12):3635-48. doi: 10.1093/brain/awq267. Epub 2010 Oct 5. PMID 20926368